CLINICAL TRIAL: NCT00713362
Title: Comparison of Chest Tube Drainage Versus Thoracoscopic Surgery for Unsuccessful Aspiration of Primary Spontaneous Pneumothorax: a Prospective Randomized Trial
Brief Title: Chest Tube Drainage or Thoracoscopic Surgery for Failed Aspiration of Spontaneous Pneumothorax
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200801030R
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-11

CONDITIONS: Pneumothorax
Keywords: Aspiration, chest tube, pneumothorax, thoracoscopic surgery
MeSH Terms: conditions — Pneumothorax | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Surgery: Video-assisted thoracoscopic surgery
  Interventions: Procedure: Video-assisted thoracoscopic surgery
- 2 (Active Comparator): Chest tube drainage
  Interventions: Procedure: chest tube drainage

INTERVENTIONS:
Procedure: Video-assisted thoracoscopic surgery — VATS for bullectomy and mechanical pleurodesis
  Arms: 1
Procedure: chest tube drainage — Chest tube drainage for pneumothroax
  Arms: 2

SUMMARY:
We hypothesize that VATS is more effective than CTD for management of primary spontaneous pneumothorax with aspiration failure. To this end, we will compare two groups of patients who had experienced unsuccessful aspiration of primary spontaneous pneumothorax stratified by treatment.

DETAILED DESCRIPTION:
Primary spontaneous pneumothorax most commonly occurs in young, tall, lean males [1, 2]. Optimal management for a first episode of this benign disease has been a matter of debate. In the recently published BTS guidelines [3], simple aspiration is recommended as the first-line treatment for all primary pneumothoraces requiring intervention because it appears to be as effective as chest tube drainage (CTD), as well as safe, well tolerated and feasible in an outpatient setting in the majority of cases [3]. When simple aspiration was unsuccessful, which occurred in about 15-62% of all pneumothoraces requiring intervention, chest tube drainage is recommended [3-12]. However, many prospective studies that have compared simple aspiration and tube drainage for primary spontaneous pneumothorax have shown that they are equally effective for treatment of primary spontaneous pneumothorax in terms of success and recurrence rates [4, 11, 12]. In this regard, chest tube drainage provides no benefits in unsuccessful aspiration of primary spontaneous pneumothorax because the rates of persistent air leakage and recurrence remain the same.

Advances in video-assisted thoracoscopic surgery (VATS) have made it a safe, less-invasive and more-effective intervention for treating recurrent pneumothorax or persistent air leakage after CTD [13-15]. However, the role of VATS in the management of first primary spontaneous pneumothorax where aspiration has failed remains unclear. Theoretically, unsuccessful aspiration is usually associated with large or persistent air leaks. Definitive treatment would include elimination of air leakage and, if possible, recurrence. Under such consideration, VATS with bullectomy and mechanical pleurodesis provides a good alternative in terms of achieving these therapeutic goals. We hypothesize that VATS is more effective than CTD for management of primary spontaneous pneumothorax with aspiration failure. To this end, we will compare two groups of patients who had experienced unsuccessful aspiration of primary spontaneous pneumothorax stratified by treatment.

This study will be performed at National Taiwan University Hospital (40 patients), Far-Eastern Memorial Hospital (10 patients), and Min-Sheng General Hospital (10 patients). A total of 60 patients will be included (30 patients in each arm).

References:

1. Gobbel WG Jr, Rhea WG, Nelson IA, Daniel RA Jr. Spontaneous pneumothorax. J Thorac Cardiovasc Surg 1963;46:331-45.
2. Lichter J, Gwynne JF. Spontaneous pneumothorax in young subjects. Thorax 1971;25:409-17.
3. Henry M, Arnold T, Harvey J. Pleural Diseases Group, Standards of Care Committee, British Thoracic Society. BTS guidelines for the management of spontaneous pneumothorax. Thorax 2003;58 (Suppl 2):39-52.
4. Harvey J, Prescott RJ. Simple aspiration versus intercostal tube drainage for spontaneous pneumothorax in patients with normal lungs. British Thoracic Society Research Committee. BMJ 1994;309:1338-9.
5. Packham S, Jaiswal P. Spontaneous pneumothorax: use of aspiration and outcomes of management by respiratory and general physicians. Postgrad Med J 2003;79:345-7.
6. Chan SS, Lam PK. Simple aspiration as initial treatment for primary spontaneous pneumothorax: Results of 91 consecutive cases. J Emerg Med 2005;28:133-8.
7. Mendis D, El-Shanawany T, Mathur A, Redington AE. Management of spontaneous pneumothorax: are British Thoracic Society guidelines being followed? Postgrad Med J 2002;78:80-4.
8. Ng AW, Chan KW, Lee SK. Simple aspiration of pneumothorax. Singapore Med J 1994;35:50-2.
9. Markos J, McConigle P, Phillips MJ. Pneumothorax: treatment by small-lumen catheter aspiration. Aust NZ J Med 1990;20:775-81.
10. Andrivet P, Djedaini K, Teboul JL, Brochard L, Dreyfuss D. Spontaneous pneumothorax. Comparison of thoracic drainage vs immediate or delayed needle aspiration. Chest 1995;108:335-40.
11. Noppen M, Alexander P, Driesen P, Slabbynck H, Verstraeten A. Manual aspiration versus chest tube drainage in first episodes of primary spontaneous pneumothorax: a multicenter, prospective, randomized pilot study. Am J Respir Crit Care Med 2002;165:1240-4.
12. Ayed AK, Chandrasekaran C, Sukumar M. Aspiration versus tube drainage in primary spontaneous pneumothorax: a randomized study. Eur Respir J 2006;27:477-82.
13. Baumann MH, Strange C, Heffner JE, Light R, Kirby TJ, Klein J, Luketich JD, Panacek EA, Sahn SA. AACP Pneumothorax Consensus Group. Management of spontaneous pneumothorax: an American College of Chest Physicians Delphi consensus statement. Chest 2001;119:590-602.
14. Naunheim KS, Mack MJ, Hazelrigg SR, Ferguson MK, Ferson PF, Boley TM, Landreneau RJ. Safety and efficacy of video-assisted thoracic surgical techniques for the treatment of spontaneous pneumothorax. J Thorac Cardiovasc Surg 1995;109:1198-204.
15. Mouroux J, Elkaim D, Padovani B, Myx A, Perrin C, Rotomondo C, Chavaillon JM, Blaive B, Richelme H. Video-assisted thoracoscopic treatment of spontaneous pneumothorax: technique and results of one hundred cases. J Thorac Cardiovasc Surg 1996;112:385-91.
16. Chen JS, Hsu, HH, Kuo SW, Tsai PR, Chen RJ, Lee JM, Lee YC. Needlescopic versus conventional video-assisted thoracoscopic surgery for primary spontaneous pneumothorax: a comparative study. Ann Thorac Surg 2003;75:1080-5.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 15 and 50 years old.
2. First episode of spontaneous pneumothorax.
3. The rim of air is > 2cm on CXR requiring simple aspiration
4. Aspiration as the initial treatment
5. Failed to achieve lung expansion following repeat manual aspiration

Exclusion Criteria:

1. Complete or nearly complete and persistent lung expansion immediately following manual aspiration
2. With underlying pulmonary disease (TB, asthma, etc)
3. With hemothorax or tension pneumothorax requiring chest tube insertion or operation
4. A history of previous pneumothorax
5. A history of previous ipsilateral thoracic operation
6. Pregnant or lactation female

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-04; Primary Completion 2012-11 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Comparing the number of days in hospital, after intervention, of each group. | within one month

SECONDARY OUTCOMES:
Short-term outcome, including number of days with chest drainage, total hospital stay, short-term failure rate of assigned treatment, adverse events, pain score, mean dose of meperidine requested. | within one month
Long-term outcome, including recurrence rate and long-term failure rate of assigned treatment | 2 years
Total costs of each patients in assigned treatment. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Chie Lee, MD, PhD, Study Chair — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei County